CLINICAL TRIAL: NCT02701166
Title: The Effect of Bezafibrate on Cholestatic Itch
Acronym: FITCH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other); University Medical Center Groningen (Other); Leiden University Medical Center (Other); UMC Utrecht (Other); Radboud University Medical Center (Other); Maastricht University Medical Center (Other); Free University Medical Center (Other); University of Barcelona (Other); Ludwig-Maximilians - University of Munich (Other); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Ruth Bolier, prof. dr. Ulrich Beuers, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL48885.018.15
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Primary Biliary Cholangitis; Primary Sclerosing Cholangitis; Secondary Sclerosing Cholangitis
Keywords: Pruritus; itch; cholestasis
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Cholangitis, Sclerosing; Pruritus; Cholestasis | interventions — Bezafibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bezafibrate (Experimental): Bezalip retard 400mg tablet
  Interventions: Drug: Bezafibrate
- Placebo (Placebo Comparator): Placebo 400mg tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bezafibrate — bezafibrate 400mg per day
  Other Names: bezalip
  Arms: Bezafibrate
Drug: Placebo — placebo 400mg per day
  Arms: Placebo

SUMMARY:
Randomized double blind placebo controlled trial to evaluate the antipruritic effect of bezafibrate in patients with moderate to severe cholestatic itch.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary biliary cholangitis or primary/secondary sclerosing cholangitis as defined by EASL clinical practice guidelines of cholestasis 2009;
* itch without primary dermatologic abnormalities and with an intensity score of ≥ 5.0 cm on a scale from 0.0 cm (no itch) to 10.0 cm (worst itch possible), scored twice in the week before inclusion.

Exclusion Criteria:

* Concomitant guideline-recommended as well as experimental antipruritic therapy, e.g.

rifampicin, opioid-receptor antagonists (naltrexon, naloxone), serotonin-reuptake inhibitors (sertraline), ondansetron, phenobarbital, propofol, lidocaine, dronabinol, butorphanol, internal or external biliary drainage, extracorporeal albumin dialysis, ultraviolet-B phototherapy; NB. Topical menthol containing agents are allowed, as well as bile salt sequestrants (colesevelam, cholestyramin) as long as taken at least 4 hours before or after intake of the study medication. Incidental use of these agents should be noted by patients in the diary, structural use should be noted on the CRF (section co-medication);

* Pregnancy, women of childbearing potential not using contraception, breast feeding;
* Cholestasis due to obstruction that requires invasive desobstructive treatment within the time scope of the study (5 weeks), such as endoscopic retrograde cholangiopancreaticography (ERCP) or surgical removal of a tumor compressing the bile duct;
* Use of opiates;
* Renal insufficiency (creatinine clearance <60mL/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a reduction in itch intensity of 50% or more | 3 weeks

SECONDARY OUTCOMES:
Serum liver tests | 3 weeks
Serum creatinine | 3 weeks
Serum cholesterol | 3 weeks
Serum autotaxin activity | 3 weeks
Serum creatinin kinase | 3 weeks

CONTACTS AND LOCATIONS:
Locations (9):
- Netherlands (8):
  - Academic Medical Center, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- University of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Vries E, Bolier R, Goet J, Pares A, Verbeek J, de Vree M, Drenth J, van Erpecum K, van Nieuwkerk K, van der Heide F, Mostafavi N, Helder J, Ponsioen C, Oude Elferink R, van Buuren H, Beuers U; Netherlands Association for the Study of the Liver-Cholestasis Working Group. Fibrates for Itch (FITCH) in Fibrosing Cholangiopathies: A Double-Blind, Randomized, Placebo-Controlled Trial. Gastroenterology. 2021 Feb;160(3):734-743.e6. doi: 10.1053/j.gastro.2020.10.001. Epub 2020 Oct 5. PMID 33031833
- [Derived] Bolier R, de Vries ES, Pares A, Helder J, Kemper EM, Zwinderman K, Elferink RPO, Beuers U; Netherlands Association for the Study of the Liver (NASL) Cholestatic Liver Diseases Study Group. Fibrates for the treatment of cholestatic itch (FITCH): study protocol for a randomized controlled trial. Trials. 2017 May 23;18(1):230. doi: 10.1186/s13063-017-1966-8. PMID 28535810